CLINICAL TRIAL: NCT06653881
Title: Comparison of Conventional and Cu-NiTi Archwires Regarding Clinical Efficiency and Pain Intensity Using Prostaglandin E2 Biomarker During Alignment and Levelling: a Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAGHAVI V
Record Dates: First submitted 2024-06-08; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Anterior Teeth Alignment Efficiency; Pain Perception; PGE2 Biomarker and Their Correlation
Keywords: TEETH ALIGNMENT; PGE2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1: Patient receiving 0.016" A-NiTi (Conventional)archwire. (Experimental): Pretreament orthodontic records (T0) of all the patients undergoing study will be taken before bonding. Before bonding, teeth will be isolated and oral prophylaxis will be performed. Enamel will be etched with 37% phosphoric acid gel, rinsed with water and air dried till a frosty appearance of the etched surface was evident. Bonding agent will be applied and cured using LED curing light unit. A conventional orthodontic adhesive will be used to bond brackets with 0.022 ̎×0.028 inch slot. In this group ,1 0.016"A-NiTi initial archwire will be securely ligated .
  Interventions: Other: ARCHWIRE
- GROUP 2:Patient receiving 0.016" Cu-NiTi archwire. (Experimental): . Pretreament orthodontic records (T0) of all the patients undergoing study will be taken before bonding. Before bonding, teeth will be isolated and oral prophylaxis will be performed. Enamel will be etched with 37% phosphoric acid gel, rinsed with water and air dried till a frosty appearance of the etched surface was evident. Bonding agent will be applied and cured using LED curing light unit. A conventional orthodontic adhesive will be used to bond brackets with 0.022 ̎×0.028 inch slot. In this group 0.016" Cu-NiTi archwire will be securely ligated.
  Interventions: Other: ARCHWIRE

INTERVENTIONS:
Other: ARCHWIRE — Alignment efficiency of the archwires will be compared using little's irregularity index between the two groups

SUMMARY:
Orthodontic treatment can inflame the periodontium and dental pulp, it can be uncomfortable and even painful at times. This may induce discomfort and the release of different biochemical mediators, which is one of the main causes of apprehension and the thing people detest the most before getting orthodontic treatment[1]. The gingival crevicular fluid (GCF), which surrounds the teeth, may exhibit particular chemical levels that indicate an inflammatory reaction that may occur throughout the orthodontic treatment procedureThe inflammatory response that arises during orthodontic treatment is mediated mostly by prostaglandin E2 (PGE2). Bone resorption may result from PGE2's activation of osteoclastic cells and increases vascular dilatation and permeability.Both rats and humans showed increased tooth movement when local prostaglandins were administered subperiosteally injected..Osteoclastic activity occurs on the pressure side of a tooth in response to an external stimulus. Simultaneously, the growth and maturation of mesenchymal stem cells (MSCs) and periodontal ligament (PDL) fibroblasts promote greater bone formation by osteoblasts on the tension side. Additionally, in osteoblasts, mechanical stress rapidly starts several cellsignalingpathways, such as those for calcium (Ca2+), nitric oxide (NO), interleukin-1 (IL-1), and adenosine triphosphate (ATP).PGE2 secretion, ATP release, and osteoblast growth are all caused by fluid shear stress activating the Ca2+ signaling pathway. The PDL experiences reduced blood flow and hypoxia at the same time on the compression side. As a result of the transcription factor HIF-1, PDL fibroblasts, and osteoblasts express VEGF and RANK-L, which stimulates osteoclast development and bone resorption in compression zones. As orthodontic movement occurs, this link becomes apparent when the alveolar bone around the tooth's root is remodelled[2]. Pain is a common side effect of orthodontic therapy, which can be very concerning to patients. Up to 72 to 100% of patients report feeling some degree of discomfort during orthodontic treatment, suggesting that many people believe the procedure to be quite painful. Unfortunately, this dread of discomfort might keep some people from ever pursuing orthodontic treatment, and it can even lead to others stopping their treatment after it has begun. Orthodontic discomfort can be effectively measured with the visual analog scale; however, its subjective character may have certain limitations. To select the most appropriate and successful type of archwires, the orthodontist must be aware of the distinctive qualities of each kind that is offered. The prevalence of stainless-steel wires for first alignment has declined with the development of nickel-titanium (NiTi) archwires.A material that can be produced stably to stop phase transition is nickel-titanium (NiTi) alloy. Additionally, it can exist in an active form with two different crystalline or lattice structures, called the austenitic (A) and martensitic (M) forms, each having specific mechanical and physical properties. The application of stress or a temperature change can cause the wire to transition between these two phases, changing its properties without compromising its structural integrity[4]. Wires have a remarkable phenomenon known as superelasticity, which is also called plateau behavior. These wires are very useful, especially for initial aligning archwires, because they can exert constant forces regardless of the degree of bending. The transition temperature, which may be predicted during the production process, is the temperature at which an alloy changes from one phase to another. Compared to other archwires, the A-NiTi archwire has exceptional spring-back characteristics. It is usual practice to add copper (Cu) to nickel-titanium (NiTi) alloy. The purpose of this adjustment is to lessen loading stress and offer the ideal force for efficient orthodontic tooth movement. Based on its phase transition and temperature dependency, the Cu-NiTi archwire displays thermo-elastic characteristics. In best of my knowledge there is no any study who had compared the effect of two wires using PGE2 levels at different intervals in levelling and alignment. This study will compare the clinical outcomes of orthodontic treatment using NiTi against Cu-NiTi archwires in terms of tooth alignment rate and pain threshold by PGE2 biomarker.

DETAILED DESCRIPTION:
Title: Comparison of conventional and Cu-NiTi archwires regarding clinical efficiency and pain intensity using prostaglandin E2 biomarker during alignment and levelling: a randomized clinical trial" Rationale:An initial archwire should be effective in aligning the arches while resulting in minimal pain and root resorption. An ideal aligning archwire should have good formability, spring back, stiffness biocompatibility, low friction, and joinability and of low cost. Orthodontic force when exerted on teeth, activates the sensory receptors in periodontal tissues and results in a nociceptive impulse processing in both the central and peripheral nervous systems. A cascade of self-limiting inflammatory reactions including cellular, vascular, neural, and immunological reactions comes into act. In particular, the locally released prostaglandin binds to the periodontal sensory endings which generates a painful sensation resulting in orthodontic pain and tooth movement. PGE2, a cyclooxygenase product, is the best-known lipid mediator that contributes to pain. Thus, the evaluation of PGE2 concentration in GCF would provide an accurate and site-specific insight on objective pain. Furthermore, the VAS score will provide knowledge of the subjective pain perceived by the patients during the initial arch- wire placement.

Therefore, it is important to assess the time point at which the patient undergoing fixed orthodontic treatment will have the maximum pain and therefore in requirement of an analgesic. This is of particular concern during the initiation of treatment since the pain would be compounded with the natural anxiety associated with the orthodontic treatment.

Aims and Objectives: To determine and compare the alignment efficiency and pain perception of 0.016" A-NiTi vs 0.016" Cu-NiTi over 12 weeks period.

Setting: Department of Orthodontics and DentofacialOrthopaedics, PGIDS, Rohtak Study Design:Two-arm parallel single-blind randomized clinical trial. Time frame: 12 weeks after initial archwire placement.

Population/participant:

Inclusion criteria:-Orthodontic patients to be treated with fixed orthodontic treatment requiring non-extraction treatment plan, moderate crowding between 4-6mm in the mandibular anterior region, between 18 and 25 years of age with full complement of teeth erupted to the occlusal level (excluding third molars)optimal periodontal condition and good oral hygiene.

Exclusion Criteria:- craniofacial anomalies and syndromes, congenitally missing teeth (excluding third molars) or severe facial asymmetries ,any systemic disease affecting bone and general growth ,acute or chronic medical patients that are under medications and would affect tooth movement, known allergy to metal and components used in orthodontic treatment.

Sample size:The sample size for the proposed study was calculated by using the formula. Total sample size = N = 2σ2(Zβ+ Zα/2) 2 / (difference)2. A sample size of 13 patients was calculated by using the above formula at confidence interval 95% with power 80%. Accounting for a 10% drop out rate, 15 patients will be enrolled in each group.

Method of study: Pre- treatment records will be taken will be selected from patients reporting to the Department of Orthodontics and Dentofacial Orthopedics, PGIDS, Rohtak. Subjects satisfying inclusion criteria will be divided into two groups.

Group 1 (G1) 0.016"A-NiTi - In this group, pretreament orthodontic records (T0) of all the patients undergoing study will be taken before bonding. Before bonding, teeth will be isolated and oral prophylaxis will be performed. Enamel will be etched with 37% phosphoric acid gel, rinsed with water and air dried till a frosty appearance of the etched surface was evident. Bonding agent will be applied and cured using LED curing light unit. A conventional orthodontic adhesive will be used to bond brackets with 0.022 ̎×0.028 inch slot. 0.016"A-NiTi initial archwire will be securely ligated with elastomeric modules.

Group 2 (G2) 0.016" Cu-NiTi-In this group, pretreament orthodontic records (T0) of all the patients undergoing study will be taken before bonding. Before bonding, teeth will be isolated and oral prophylaxis will be performed. Enamel will be etched with 37% phosphoric acid gel, rinsed with water and air dried till a frosty appearance of the etched surface was evident. Bonding agent will be applied and cured using LED curing light unit. A conventional orthodontic adhesive will be used to bond brackets with 0.022 ̎×0.028 inch slot. 0.016" Cu-NiTi archwire will be securely ligated with elastomeric modules.

Outcome Measures: Changes in the following parameters -little's irregularity index will be measured by model scanning in both the groups. Assessment of these parameters will be done at T0 (baseline data), T1(6 weeks after initial archwire placement), T2(12 weeks after initial archwire placement). Gingival crevicular fluid (GCF) will be collected 1 hr before bonding in lower arch , 24 hours after initial arch wire placement , 48 hrs after initial arch wire placement , 72hrs after initial arch wire placement for assessing PGE2 levels. Pain assessment will be done at 24 hours after initial archwire placement, 48 hours after initial archwire placement, 72 hours after initial archwire placement.

Statistical Analysis: Descriptive statistics and inferential statistics will be used. Data will be checked for normality. In all the analysis, the level of significance will be set at 5 percent.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients to be treated with fixed orthodontic treatment requiring non-extraction treatment plan.
* Patients' with pre-treatment moderate crowding between 4-6mm in the mandibular anterior region assessed with Little's Irregularity index.
* Male and female patients between 18 and 25 years of age with full complement of teeth erupted to the occlusal level (excluding third molars).
* Non syndromic patients and no impaction of teeth except third molars.
* No history of previous orthodontic treatment.
* Optimal periodontal condition and good oral hygiene.

Exclusion Criteria:

* Acute or chronic medical patients that are under medications and would affect tooth movement.
* Medical conditions that contraindicate orthodontic treatment.
* Craniofacial anomalies and syndromes, congenitally missing teeth (excluding third molars) or severe facial asymmetries.
* Any systemic disease affecting bone and general growth.
* Patients' with known allergy to metal and components used in orthodontic treatment.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
ARCH ALIGNMENT | T0 - Baseline records, at the time before treatment
  compare anterior teeth alignment efficiency with little's irregularity index in 'mm' using cast scanning with meshlab software
ARCH ALIGNMENT | T1 - Records at 6th week after wire placement
  compare anterior teeth alignment efficiency with little's irregularity index in 'mm' using cast scanning with meshlab software
ARCH ALIGNMENT | T2 - Records at 12th week after wire placement
  compare anterior teeth alignment efficiency with little's irregularity index in 'mm' using cast scanning with meshlab software

SECONDARY OUTCOMES:
SUBJECTIVE PAIN ASSESSMENT BY VISUAL ANALOG SCALE | 1. 24 hours after initial archwire placement.
  The intensity of pain perceived by the patients will be assessed with the help of VAS score. A 100 mm VAS with scores of 0 to 10 was given with 0 meaning no pain and while 10 meant very painful
SUBJECTIVE PAIN ASSESSMENT BY VISUAL ANALOG SCALE | 2. 48 hours after initial arch wire placement
  The intensity of pain perceived by the patients will be assessed with the help of VAS score. A 100 mm VAS with scores of 0 to 10 was given with 0 meaning no pain and while 10 meant very painful.Pain assessment will be done at following time intervals
SUBJECTIVE PAIN ASSESSMENT BY VISUAL ANALOG SCALE | 3. 72 hours after initial arch wire placement
  The intensity of pain perceived by the patients will be assessed with the help of VAS score. A 100 mm VAS with scores of 0 to 10 was given with 0 meaning no pain and while 10 meant very painful.Pain assessment will be done at following time intervals

OTHER OUTCOMES:
GCF COLLECTION | 1. 1 hour before bonding in lower arch
  A sterile standardized PERIOPAPER strip will be gently inserted into the periodontal pocket/gingival sulcus until mild resistance will be felt in an attempt to minimize the mechanical trauma of gingival tissues. The collected GCF will be stored in sterile vials containing 100 μl of phosphate buffer solution. The samples will bethen centrifuged at 1000 rotations per minute for 15 minutes to settle the particulate matter.For processing, a Human PGE2 ELISA Kit will be used.
GCF COLLECTION | 2. 24hours after initial arch wire placement
  A sterile standardized PERIOPAPER strip will be gently inserted into the periodontal pocket/gingival sulcus until mild resistance will be felt in an attempt to minimize the mechanical trauma of gingival tissues. The collected GCF will be stored in sterile vials containing 100 μl of phosphate buffer solution. The samples will bethen centrifuged at 1000 rotations per minute for 15 minutes to settle the particulate matter.For processing, a Human PGE2 ELISA Kit will be used.
GCF COLLECTION | 3. 48 hours after initial arch wire placement
  A sterile standardized PERIOPAPER strip will be gently inserted into the periodontal pocket/gingival sulcus until mild resistance will be felt in an attempt to minimize the mechanical trauma of gingival tissues. The collected GCF will be stored in sterile vials containing 100 μl of phosphate buffer solution. The samples will bethen centrifuged at 1000 rotations per minute for 15 minutes to settle the particulate matter.For processing, a Human PGE2 ELISA Kit will be used.
GCF COLLECTION | 4. 72 hours after initial arch wire placement
  A sterile standardized PERIOPAPER strip will be gently inserted into the periodontal pocket/gingival sulcus until mild resistance will be felt in an attempt to minimize the mechanical trauma of gingival tissues. The collected GCF will be stored in sterile vials containing 100 μl of phosphate buffer solution. The samples will bethen centrifuged at 1000 rotations per minute for 15 minutes to settle the particulate matter.For processing, a Human PGE2 ELISA Kit will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No